CLINICAL TRIAL: NCT06703489
Title: Safety and Performance Assessment of the Sphere-9™ Catheter and Affera™ Ablation System for the Treatment of Ventricular Tachycardia
Brief Title: Safety and Performance Assessment of the Sphere-9™ Catheter and Affera™ Ablation System for the Treatment of Ventricular Tachycardia (Sphere-9 VT EFS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Ablation Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sphere-9 VT EFS
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Ventricular Tachycardia (VT)
Keywords: Recurrent sustained monomorphic ventricular tachycardia; Monomorphic ventricular tachycardia; Ventricular tachycardia; Arrhythmias, Cardiac; Heart Diseases; Cardiovascular Diseases; Pathologic Processes; Ischemic heart disease; Patient with Implantable Cardioverter Defibrillator (ICD); Ischemic cardiomyopathy
MeSH Terms: conditions — Tachycardia, Ventricular; Arrhythmias, Cardiac; Heart Diseases; Cardiovascular Diseases; Pathologic Processes; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Ventricular tachycardia catheter ablation (Experimental): Ablation using the Sphere-9 Catheter with the Affera Mapping and Ablation System
  Interventions: Device: Sphere-9 Catheter with the Affera Mapping and Ablation System

INTERVENTIONS:
Device: Sphere-9 Catheter with the Affera Mapping and Ablation System — Adult subjects with recurrent, sustained, scar-related monomorphic ventricular tachycardia will be enrolled and undergo ablation with the Sphere-9 Catheter with the Affera Mapping and Ablation System.

SUMMARY:
Sphere-9 VT EFS is a prospective, multi-center, non-randomized, unblinded feasibility study. Adult subjects with recurrent, sustained, scar-related monomorphic ventricular tachycardia will be enrolled and treated with the Sphere-9 Catheter and Affera Ablation System.

ELIGIBILITY:
Inclusion Criteria:

1. Any of the following:

   1. Ischemic cardiomyopathy (ICM) patients with prior history of myocardial infarction (MI).
   2. Non-ischemic cardiomyopathy (NICM) patients with documented myocardial scar in a territory without coronary stenosis as evidenced by cardiac imaging.
2. At least one episode of sustained (continuous for >30 seconds or requiring ICD intervention for termination) monomorphic ventricular tachycardia within the 6 months prior to enrollment.
3. Recurrence of sustained ventricular tachycardia despite class I or III antiarrhythmic drug therapy or ICD intervention.
4. Implanted with an implantable cardiac defibrillator (ICD) or CRT-D for at least 3 months prior to the ablation procedure.
5. Age 18 through 85 years old.
6. Willing and able to provide informed consent.
7. Willing and able to comply with all pre-, post-, and follow-up testing requirements.

Exclusion Criteria:

1. Incessant VT necessitating hemodynamic support prior to the ablation procedure.
2. Unstable polymorphic VT or ventricular fibrillation (VF).
3. VTs due to any of the following:

   1. Idiopathic VT
   2. Automaticity or triggered activity
   3. Lamin or titin genetic mutation
   4. Ventricular tachycardia secondary to electrolyte imbalance, active thyroid disease, or any other reversible or non-cardiac cause (e.g., drug induced arrhythmia).
4. NICM subjects with active inflammatory processes (e.g., myocarditis) within 120 days prior to the ablation procedure.
5. VT or VF thought to be from channelopathies.
6. More than two prior VT ablations at any time, more than one prior VT ablation within 12 months prior to the ablation procedure, or any VT ablation within 4 weeks prior to the ablation procedure.
7. Sarcoidosis.
8. Hypertrophic cardiomyopathy, except when due to an apical aneurysm.
9. Unstable angina.
10. Active myocardial ischemia.
11. Type 1 myocardial infarction within 2 months (60 days) prior to the ablation procedure.
12. Any percutaneous coronary intervention within 2 months (60 days) prior to the ablation procedure.
13. Any cardiac surgery within 3 months (90 days) prior to the ablation procedure.
14. Left ventricular ejection fraction (LVEF) <15%.
15. NYHA Class IV heart failure.
16. Decompensated heart failure.
17. Currently receiving support, or anticipated to receive support prior to the index ablation procedure, via extracorporeal membrane oxygenation (ECMO).
18. Ventricular assist device (VAD) implanted, planned or required for the procedure.
19. Severe aortic or mitral stenosis, or severe aortic or mitral regurgitation.
20. Presence of prosthetic valve in the aortic or mitral valve.
21. Patients with advanced COPD (on home oxygen).
22. Presence of intracardiac thrombus, tumor, or other abnormality that precludes vascular access, catheter introduction, or manipulation.
23. Thromboembolic event (stroke or transient ischemic attack) within 6 months (180 days) prior to the index ablation procedure or with neurologic deficit.
24. Left atrium (LA) or left ventricle (LV) intracardiac thrombus on imaging.
25. Severe bleeding, clotting or thrombotic disorder, or thrombocytopenia (defined as platelet count <80,000).
26. Contraindication to anticoagulation.
27. End-stage renal disease (requiring dialysis).
28. Acute illness, active infection, or sepsis.
29. Life expectancy less than 12 months.
30. Any woman known to be pregnant or breastfeeding, or any woman of childbearing potential who is not on a reliable form of birth regulation method or abstinence.
31. Body mass index >45 kg/m2.
32. Known ongoing drug or alcohol dependency.
33. Current or anticipated participation in any other ongoing study of a drug, device, or biologic during the duration of the study not pre-approved by the Sponsor.
34. Vulnerable subjects (such as a prisoner, handicapped or mentally disabled person, or person under tutelage or guardianship).
35. Any other condition that, in the opinion of the investigator, would preclude enrollment in this study or compliance with follow-up requirements or would pose a significant hazard to the subject if an ablation procedure were performed.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint: evaluate the safety of the index ablation procedure | Within 7 days post-procedure
  Percentage of patients with device- or procedure-related cardiovascular- or pulmonary-related serious adverse events
Primary Effectiveness Endpoint: assess acute procedural success of the index ablation procedure | Day of ablation procedure
  Percentage of patients whose targeted clinically relevant monomorphic ventricular tachycardia cannot be induced

SECONDARY OUTCOMES:
Secondary Endpoint: assess chronic effectiveness of the index ablation procedure | Within 6 months post-procedure
  Percentage of patients free from recurrence of sustained monomorphic ventricular tachycardia

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (5):
- United States (5):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No